CLINICAL TRIAL: NCT06615206
Title: An Open-label, Multiple-dose Clinical Study to Evaluating the Safety, Tolerability and Preliminary Efficacy of a Single Intracerebroventricular Injection of HG204 for the Treatment of MECP2 Duplication Syndrome
Brief Title: A First-in-Human Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of a Novel CRISPR RNA-editing Therapy in Patients with Mecp2 Duplication Syndrome, a Rare Orphan Disease (HERO)
Acronym: HERO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HuidaGene Therapeutics Co., Ltd. (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HG20401
Record Dates: First submitted 2024-09-04; First posted 2024-09-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: MECP2 Duplication Syndrome
Keywords: MECP2; dupMECP2; CNS; neurodevelopmental disease; Gene-editing; HG204; CRISPR; MDS
MeSH Terms: conditions — Lubs X-linked mental retardation syndrome

STUDY DESIGN:
Intervention Model Description: Open-label, multiple doses of a single intracerebroventricular injection of HG204
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HG204 (Experimental): Once intracerebroventricular injection; The duration of the study is about 60 weeks for each subject, including a 8 weeks screening period, enrollment visit, treatment visit and 52 weeks follow-up period.
  Interventions: Genetic: HG204

INTERVENTIONS:
Genetic: HG204 — The study will enroll up to 2 cohorts, evaluating a starting dose plus a higher or lower dose

SUMMARY:
Methyl-CpG binding protein 2 (MECP2) is a dosage-sensitive, X-linked gene critical for central nervous system development and functional maintenance, which gain-of-function causes MECP2 duplication syndrome (MDS). Affecting primarily in males, this disorder is characterized by severe intellectual disability, motor dysfunction, infantile hypotonia, epilepsy, respiratory tract infections, and premature death before 25 years of age with no curative therapy.

HG204 is a CRISPR RNA-editing therapy packaging novel high-fidelity Cas13Y (hfCas13Y) technology, using one single adeno-associated virus (AAV) vector to target and knock down MECP2 mRNA in the brain. Preclinical studies showed that a single intracerebroventricular injection of HG204 persistently decreased MECP2 mRNA and MECP2 protein in the cortex of the MDS mice, reversed the abnormal motor and social phenotypes, and significantly prolonged survival in MDS mouse models.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 2 and ≤18 years at the time of signing informed consent;
* Genetic test and clinical confirmed diagnosis of MDS;
* Stable pattern of seizures, or has had no seizures while currently receiving medical treatment (including antiepileptics) and physical therapy are stable for at least 2 months before screening;
* Willing to adhere to protocol, including biological samples collection and hospitalization for intracerebroventricular injection surgery;
* Acceptable hematology, clinical chemistry, and urine laboratory parameters.

Exclusion Criteria:

* MECP2 gene triplication;
* Concurrent genetic syndromes other than MDS;
* Significant brain or cerebellar atrophy, or other significant degenerative changes as shown in cranial MRI at screening;
* Prior or current hypertension, cardiomyopathy, myocardial ischemia or atrial fibrillation and other cardiovascular diseases;
* Prior central nervous system surgery within 6 months before enrolment;
* Systemic use of immunosuppressive drugs within 3 months before enrolment;
* Prior gene therapy or oligonucleotide therapy treatments;
* Any other conditions that would not allow the potential subject to complete follow-up examinations during the study and would, in the opinion of the investigator, make the potential subject unsuitable for the study.

Ages: 2 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of systemic adverse events | 52 weeks
  Number of adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impression Scale | 52 weeks
  Clinical Global Impression Scale is a scale to evaluate mental disorder severity, with a score range from 1-7, the higher scrore means worse mental disorder.
Change from baseline in Griffiths Developmental Assessment Scale | 52 weeks
  Griffiths Developmental Assessment Scale is a scale to evaluate mental development function of children aged 0-8, including sensory, cognitive and movement, the minimum score is 0, and no maximum limit for the highest score, the higher score means better mental development.
Change from baseline in Peabody Developmental Assessment Scale | 52 weeks
  Peabody Developmental Assessment Scale is a scale to evaluate motor function of children aged 0-6, with a score range from 0-100, the higher scrore means better motor function.
Change from baseline in Wechsler (toddler/child) Intelligence Scale (fourth version) score | 52 weeks
  Wechsler (toddler/child) Intelligence Scale (fourth version) score is a scale to assessing the intelligence of children aged 6 to 16, the score range showed a normal distribution, there is no minimum and maximum score, score from 90 to 110 points is normal intelligence result, the higher score means better intelligence.
Adaptive Behavior Rating Scale | 52 weeks
  Adaptive Behavior Rating Scale is a scale assessing daily living ability of children aged 0-18, with a score range from 0-200, the higher score means better daily living ability

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No